CLINICAL TRIAL: NCT06653036
Title: Dural Puncture Epidural Vs Standard Epidural Technique in Parturient Receiving Continuous Labour Epidural Infusion: a Randomized Controlled Trial
Brief Title: Dural Puncture Epidural Vs Standard Epidural Technique in Parturient Receiving Continuous Labour Epidural Infusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Samina Ismail, Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2024-10424-31009
Record Dates: First submitted 2024-09-26; First posted 2024-10-22 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Quality Health Care
Keywords: Quality Labor Analgesia; Maternal Adverse Events

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DPE group (Active Comparator): Participants who receive the dural puncture epidural (DPE) for labor analgesia.
  Interventions: Procedure: Dural puncture epidural
- SET group (Active Comparator): Participants who will be receiving standard epidural technique (SET) for labor analgesia.
  Interventions: Procedure: Standard Epidural Technique

INTERVENTIONS:
Procedure: Dural puncture epidural — The Dural puncture epidural technique is done by assessing the epidural space using the Touhy needle and puncturing the dura matter with a finer needle.
  Arms: DPE group
Procedure: Standard Epidural Technique — The Standard Epidural Technique is usually performed by identifying the epidural space using the loss of resistance technique and threading the epidural catheter in the epidural space for administration of analgesic drugs.
  Arms: SET group

SUMMARY:
The goal of this study is to evaluate the quality and safety of labor analgesia by comparing the use of Dural puncture epidural technique to Standard epidural technique while maintaining labor analgesia by means of continuous epidural infusion in parturient. The main questions it aims to answer are

* Effectiveness and quality of labor analgesia
* Frequency of catheter adjustments
* Need for catheter replacements
* Incidence of failed regional anesthesia requiring conversion to general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous / Multiparous women
* Age >18 years
* ASA 1 & 2
* Singleton vertex presentation
* Gestational age 37-42 weeks
* Parturient with established labor and pain score ≥ 3

Exclusion Criteria:

* Major cardiac disease
* History of chronic pain
* Chronic opioid user
* Platelet count < 70 x 109/L
* spinal cord anomalies
* Use of anticoagulants
* Allergic to local anesthetics
* Patients with preeclampsia/ eclampsia
* Known fetal anomalies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | At 30 minutes of initiation of infusion
  Pain assessment by using numerical rating pain score and assessing sensory level. Numerical rating score: Pain Assessment: Numerical rating scale (NRS) 0 to 10. 0=no pain, 1-3 =mild pain, 4-7 =Moderate pain, 8-10= severe pain. Assessing sensory level: Testing will be done on specific dermatomes and will be compared bilaterally by either using one of these tests. 1. Light Touch Test: Dab a piece of cotton wool on an area of skin. 2. Temperature test: by using Ice on specific dermatomes and ask the patient if they feel cold sensation 3. Pinprick Test for pain sensation - Gently touch the skin with the pin ask the patient whether it feels sharp or blunt.
Need for catheter adjustment | At 30 minutes of initiation of infusion
  Persistence of either unilateral pain score (NRS) of >4, thirty minutes after 2 boluses of 10ml of 0.125% Bupivacaine

SECONDARY OUTCOMES:
Patient Satisfaction | At 30 minutes of initiation of infusion
  Patient Satisfaction using a five-point satisfaction score as follows:
  Satisfied (score 1 to 3) ------------- Unsatisfied (score 4 to 5) -----------
  1. perfect: the patient did not experience any pain at all,
  2. very satisfied: helped relieve most of her pains,
  3. satisfied: the epidural procedure relieved major pains, but she still experienced minor pains,
  4. 4not satisfied: the epidural procedure helped only a bit a
  5. poor: the epidural procedure did not help at all. Scores from 1 to 3 were considered as the patient being satisfied with the labour epidural analgesia, and scores from 4 to 5 were regarded as the patient being unsatisfied with the labour epidural analgesia.
Assessment of the level of motor Block | At 30 minutes after the initiation of infusion
  The level of the motor block will be assessed using the modified Bromage score. Where, 1 =unable to flex feet or knees, 2 =able to flex feet only, 3 =s able to flex knees, 4 = detectable weakness in hip flexion, 5 = no weakness with hip flexion

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No